CLINICAL TRIAL: NCT00370409
Title: Cryotherapy of Sclerotomy Sites for Prevention of Late Postvitrectomy Diabetic Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8525
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Late Postvitrectomy Diabetic Hemorrhage.
Keywords: Rebleeding; Diabetic vitreous hemorrhage; Cryotherapy
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Cryotherapy
  Interventions: Procedure: Cryotherapy
- 2 (Placebo Comparator)
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Procedure: Cryotherapy — Cryotherapy of both sides of sclerotomy sites was done for 6 seconds after complition of operation.

SUMMARY:
Late vitreous hemorrhage in postvitrectomized diabetic eyes may be due to fibrovascular tuft formation in sclerotomy sites. Cryotherapy of sclerotomy sites may prevent bleeding by regressing the fibrovascular tuft. This study will detect the safety and efficacy of cryotherapy of sclerotomy sites for prevention of late vitreous hemorrhage in vitrectomized diabetic eyes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic retinopathy cases undergoing vitrectomy

Exclusion Criteria:

* History of deep vitrectomy or cataract surgery
* Renal failure
* Silicone oil injection during surgery
* Early rebleeding
* History of antithrombotic drugs usage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Prevention of late vitreous hemorrhage in postvitrectomized diabetic eyes | 6 months

SECONDARY OUTCOMES:
Incidence of late vitreous hemorrhage in the cryo group. | 6 months
Incidence of late vitreous hemorrhage in the control group. | 6 months
Comparing incidence of late vitreous hemorrhage in both groups. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Entezari, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran